CLINICAL TRIAL: NCT00660114
Title: A Non-Interventional Study of Cough Variant Asthma Treatment With Pulmicort®Respules® in Patient Aged 5-Year Old or Younger in Outpatient Department
Brief Title: Non-Interventional Study of Cough Variant Asthma Treatment With Pulmicort®Respules® in Children Outpatients
Acronym: PUL NIS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Lars-Göran Carlsson - Medical Science Director, AstraZeneca
Other Study IDs: NIS-RCN-PUL-2008/1
Record Dates: First submitted 2008-04-15; First posted 2008-04-17 (Estimated); Last update posted 2009-05-28 (Estimated); Status verified 2009-05

CONDITIONS: Cough Variant Asthma
Keywords: Cough variant asthma; Pulmicort® Respules®; Chinese patient Eligibility
MeSH Terms: conditions — Cough-Variant Asthma

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This open label, non-interventional study is to show the efficacy of Pulmicort®Respules® in cough variant asthma in patient aged 5-year old or younger in outpatient department

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Patient who has been prescribed Pulmicort® Respules® according to physician's judgement, irrespective of the inclusion in the study.
* The usage of Pulmicort® Respules® follows local authorised package insert.

Exclusion Criteria:

* Allergy to any ingredient of Pulmicort® Respules®
* With history of Leukotriene Modifier (LM) usage prior to 2 weeks of recruitment or following plan.
* Have used systemic/inhaled steroid prior to 2 weeks of recruitment

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patient aged 5-year old or younger who has been diagnosed as cough variant asthma and decided by physician to use Pulmicort® Respules® inhalation.
Sampling Method: Non-Probability Sample
Enrollment: 914 (Actual)
Dates: Start 2008-04; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Patient Symptom Score | 7 weeks (plus or minus 3 days )

SECONDARY OUTCOMES:
Patient Compliance Report | 7 weeks (plus or minus 3 days )
Investigator Assessment Report | 7 weeks (plus or minus 3 days )

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jianguo, Professor, Principal Investigator — Shanghai Jiao Tong University Affiliated First People's Hospital
Locations (32):
- China (32):
  - Research Site, Hefei, Anhui
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Chongqing, Chongqing Municipality
  - Research Site, Quanzhou, Fujian
  - Research Site, Xiamen, Fujian
  - Research Site, Guangzhou, Guangdong
  - Research Site, Shenzhen, Guangdong
  - Research Site, Zhongshan, Guangdong
  - Research Site, Shijiazhuang, Hebei
  - Research Site, Harbin, Hei Longjiang
  - Research Site, Zhengzhou, Henan
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Changzhou, Jiangsu
  - Research Site, Nanjing, Jiangsu
  - Research Site, Suzhou, Jiangsu
  - Research Site, Wuxi, Jiangsu
  - Research Site, Nanchang, Jiangxi
  - Research Site, Changchun, Jilin
  - Research Site, Shenyang, Liaoning
  - Research Site, Jinan, Shandong
  - Research Site, Qingdao, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Taiyuan, Shanxi
  - Research Site, Xi’an, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Kunming, Yunnan
  - Research Site, Hangzhou, Zhejiang
  - Research Site, Ningbo, Zhejiang
  - Research Site, Rui’an, Zhejiang
  - Research Site, Wenzhou, Zhejiang